CLINICAL TRIAL: NCT02891369
Title: Retrospective Analysis of Patients Treated With Bevacizumab in GHPSJ Intraperitoneal for the Treatment of Refractory Malignant Ascites
Brief Title: Analysis of Patients Treated With Bevacizumab Intraperitoneal for the Treatment of Refractory Malignant Ascites
Acronym: BEVASCITE
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: BEVASCITE
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2016-09

CONDITIONS: Refractory Malignant Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention. Descriptive study

SUMMARY:
The refractory malignant ascites is a complication of advanced stages of many cancer types. It is characterized clinically by abdominal pressure sensation, shortness of breath and pelvic pain. Thus, it contributes to decreased quality of life for these patients in palliative care.

Conventional treatment is based on paracentesis of ascites. The progression of the disease leads to increased production of ascites requiring more frequent paracentesis. Main therapeutic alternatives are constituted by the controversial use of diuretics and the use of an antibody inhibiting the activity of the Vascular Endothelial Growth Factor (VEGF): bevacizumab. Catumaxomab, a monoclonal antibody anti-EpCAM and CD3, developed for the treatment of refractory malignant ascites showed no sufficient clinical benefit.

VEGF is overexpressed in many tumors. VEGF causes an increase in capillary permeability and capillary filtration surface generating increased protein extravasation. These phenomena are responsible for an increase of the volume of ascites product. Thus the use of inhibitors of VEGF, such as bevacizumab, could reduce the production of ascites.

The efficacy of bevacizumab to decrease the volume of ascites product was demonstrated on small animals in intraperitoneal administration.

Studies in humans are few and the doses used are not consistent from one study to another.

DETAILED DESCRIPTION:
Main objective / secondary:

The objective of this study is to describe the population, adverse effects, the volume of ascites product and time between paracentesis in patients receiving bevacizumab in intraperitoneal through a refractory malignant ascites.

Methodology :

This is a retrospective study mono centric and non-interventional. data collected

* Name,
* date of birth,
* dates and numbers injection of bevacizumab doses
* side effects,
* type of cancer, TNM classification,
* ascites volume collected during paracentesis prior to the introduction of IP bevacizumab,
* frequency of paracentesis before the introduction of IP bevacizumab,
* ascites volume collected during paracentesis after the introduction of IP bevacizumab,
* frequency after paracentesis after the introduction of IP bevacizumab,
* albumin
* Number of lines of chemotherapy received
* Treatment monotherapy or in combination with other chemotherapies
* WHO Stadium in each course
* Date of death

supports

* Data collection from CHIMIO® software DxCare® and non-computerized patient records.
* Series anonymized patient data on Excel®

Circulation mode and data processing and not opposition patient The anonymous data are entered on a computer file and centralized within the pharmacy department by the investigator of the Groupe Hospitalier Saint Joseph Paris, Carole METZ, to be processed locally.

For the statistical analysis, quantitative variables are expressed by their mean, standard deviations, their minimum and maximum values as appropriate. The variables will be expressed in numbers and percentages. Descriptive data analyzes, correlations between the study variables and more specific tests to determine the prognostic value of variable can be used.

This is a single-center retrospective cohort within the GHPSJ. Patients are aware of the potential use of their data in their files for medical research by information contained in the handbook of the institution for patients.

Development of the study:

* The list of patients who received bevacizumab injection is obtained from the CHIMIO® software.
* The data collected is validated by a multidisciplinary way oncologists and pharmacists.
* Collection and analysis of data by the internal pharmacy from computerized patient records (DxCare®) or not computerized.

ELIGIBILITY:
Inclusion Criteria:

* All assigns patients received at least one injection of bevacizumab intraperitoneal within GHPSJ between 01/01/2007 and 31/12/2014

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted with Refractory Malignant Ascites and wgho received bevacizumab intraperitoneal (IP) injection
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Assessment of the ascites volume | 1 Hour before introduction of bevacizumab
  Assessment of the ascites volume (mL) collected during paracentesis prior to the introduction of IP bevacizumab

SECONDARY OUTCOMES:
Assessment of the TNM classification of the cancer | Day1
  type of cancer, TNM
Assessment of the number of paracentis happened | Month 12
  frequency after paracentesis after the introduction of IP bevacizumab

CONTACTS AND LOCATIONS:
Overall Officials: Meryam JARDIN, PharmD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided